CLINICAL TRIAL: NCT02925442
Title: Comparison Between Cooled (C-RFA) and Standard (t-RFA) Radiofrequency Ablation, and Control for Pain Management Following Unilateral Knee Arthroplasty: A Double-Blinded, Parallel-Grouped, Placebo-Controlled Randomized Clinical Trial
Brief Title: Genicular Radiofrequency Ablation for Unilateral Knee Arthroplasty Pain Management
Acronym: RFA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lyman Medical Research Foundation, Inc. (Other)
Collaborators: Halyard Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OSI-0002
Record Dates: First submitted 2016-10-03; First posted 2016-10-05 (Estimated); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Osteoarthritis of the Knee
Keywords: Unilateral Knee Arthroplasty; Radiofrequency Ablation; Genicular; RFA; C-RFA; t-RFA; total knee replacement
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Genicular radiofrequency ablation performed prior to total knee arthroplasty for pain management
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Thermal radiofrequency ablation (Experimental): Patients randomized to t-RFA will receive standard genicular thermal radiofrequency ablation at least 3 weeks prior to unilateral knee arthroplasty for postoperative pain management.
  Interventions: Procedure: t-RFA
- Cooled radiofrequency ablation (Experimental): Patients randomized to C-RFA will receive cooled genicular thermal radiofrequency ablation at least 3 weeks prior to unilateral knee arthroplasty for postoperative pain management.
  Interventions: Procedure: C-RFA
- Control:Placebo Sham (Sham Comparator): Patients randomized to control will receive simulated genicular thermal radiofrequency ablation at least 3 weeks prior to unilateral knee arthroplasty and receive the industry standard of care for unilateral knee arthroplasty pain management.
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: t-RFA — standard thermal genicular radiofrequency ablation
  Other Names: Standard thermal genicular radiofrequency ablation
  Arms: Standard Thermal radiofrequency ablation
Procedure: C-RFA — Cooled radiofrequency ablation
  Other Names: Coolief radiofrequency ablation
  Arms: Cooled radiofrequency ablation
Procedure: Control — Simulated radiofrequency ablation for placebo controlled group
  Other Names: Placebo Sham
  Arms: Control:Placebo Sham

SUMMARY:
Three primary reasons prolong hospital stays following unilateral knee arthroplasty. Pain is the primary reason followed by opioid drowsiness and nausea/vomiting side effects. Standard genicular radiofrequency ablation (t-RFA) has been effective pain management for non-operative knee pain associated with osteoarthritis. Additionally, cooled radiofrequency ablation (C-RFA), is now available for knee pain management. Both t-RFA and C-RFA offer minimally invasive, non-surgical, non-opioid pain relief options following surgery. The study will perform a double-blinded, parallel grouped, placebo-controlled randomized study to compare three pain management paradigms involving preoperative genicular C-RFA, t-RFA, and control placebo/sham. The aim of this study is to establish if C-RFA and t-RFA, offered preoperatively to patients undergoing unilateral knee arthroplasty, provide postoperative pain relief.

DETAILED DESCRIPTION:
Total knee replacements are a leading orthopedic procedure in the United States totaling 600,000 in 2010, and are anticipated to grow to 3.48 million procedures by 2030. Three primary reasons prolong hospital stays following unilateral knee arthroplasty. Pain is the primary reason followed by opioid drowsiness and nausea/vomiting side effects. Reducing opioid usage and decreasing hospital length of stays are paramount in improving patient care during recovery and rehabilitation, subsequently reducing overall costs associated with total knee replacement. Standard genicular radiofrequency ablation (t-RFA) has been effective pain management for non-operative knee pain associated with osteoarthritis. Additionally, cooled radiofrequency ablation (C-RFA), which was previously used for spinal pain, is now available for knee pain management. C-RFA, compared to t-RFA, causes large volume spherical lesions and potentially reduces time and fluoroscopic exposure with direct placement techniques. However, both t-RFA and C-RFA offer a minimally invasive, non-surgical, non-opioid pain relief options following surgery. Preliminary reports involving 40 patients who underwent either C-RFA or t-RFA prior to unilateral knee arthroplasty by the investigator indicate both procedures improved postoperative pain assessments and decreased opioid/narcotic utilization. The study will perform a double-blinded, parallel grouped, placebo-controlled randomized study to compare three pain management paradigms involving preoperative C-RFA, t-RFA, and sham. The aim of this study is to establish if C-RFA and t-RFA, offered preoperatively to patients undergoing unilateral knee arthroplasty, provide postoperative pain relief, reduce hospital length of stays and decrease opioid utilization thereby improving patient outcomes and decreasing overall costs.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of the knee where unilateral knee arthroplasty is indicated by radiograph, function decrease and/or pain indication and readiness to undergo t-RFA, C-RFA or sham treatment.

Exclusion Criteria:

□ • NO DAILY OPIOID CONSUMPTION 5 WEEKS PRIOR TO ENROLLMENT

* NO DOCUMENTED NARCOTIC DEPENDENCY OR RECREATIONAL DRUG USE
* NO TOBACCO USAGE WITHIN 2 MONTHS PRIOR TO SURGERY
* NO CONFOUNDING INFLAMMATORY ARTHRITIS DISEASES ARE PRESENT
* NO NEUROPATHY OR NEURO IMPAIRMENT PRESENT
* NO SIGNIFICANT ACUTE ILLNESS OR INFECTION
* NO OTHER CONFOUNDING CHRONIC PAIN
* NO INVESTIGATIONAL AGENT WITHIN 3 MONTHS PRIOR TO ENROLLMENT
* NO DIAGNOSED THROMBOPHILIA
* NO SEVERE CARDIAC OR PULMONARY COMPROMISE
* NO BLEEDING DISORDER(S)
* NO ALLERGIC REACTION TO LOCAL ANESTHESIA, STEROIDS, OR IMPLANT MATERIALS
* NO BREASTFEEDING
* NO PREGNANCY
* NO CONFOUNDING PSYCHIATRIC ILLNESSES
* NO CONFOUNDING MAJOR TRAUMA HARDWARE REMOVALS OR PRIOR TKA *NO CONTRAINDICATED BODY HABITUS TO BE DETERMINED BY A TREATMENT PROVIDER

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-01-25 (Actual); Primary Completion 2020-01-07 (Estimated); Study Completion 2020-02-07 (Estimated)

PRIMARY OUTCOMES:
Postoperative analgesic consumption | 0 - 3 weeks postoperatively
  Measure opioid consumption for the three study arms
Hospital Length of Stay (LOS) | 0-5 days postoperatively
  Measure hospital length of stay for the three study arms

SECONDARY OUTCOMES:
Pain Score | before treatment arm procedures to 12 months after unilateral knee arthroplasty
  assess patient pain score diaries after total knee replacement for the three treatment arms

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Lyman, MD, Principal Investigator — Orthopedic Specialty Institute; Timothy Lovell, MD, Principal Investigator — Providence Medical Center
Locations (2):
- United States (2):
  - Orthopedic Specialty Institute, Coeur d'Alene, Idaho
  - Orthopedic Specialty Institute, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schiltenwolf M, Fischer C. Choi WJ et al. Radiofrequency treatment relieves chronic knee osteoarthritis pain: a double-blind randomized controlled trial. Pain 2011; 152: 481-7. Pain. 2011 Aug;152(8):1933-1934. doi: 10.1016/j.pain.2011.05.031. Epub 2011 Jun 22. No abstract available. PMID 21700390
- [Background] Husted H, Lunn TH, Troelsen A, Gaarn-Larsen L, Kristensen BB, Kehlet H. Why still in hospital after fast-track hip and knee arthroplasty? Acta Orthop. 2011 Dec;82(6):679-84. doi: 10.3109/17453674.2011.636682. Epub 2011 Nov 9. PMID 22066560
- [Background] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Background] Patel A, Pavlou G, Mujica-Mota RE, Toms AD. The epidemiology of revision total knee and hip arthroplasty in England and Wales: a comparative analysis with projections for the United States. A study using the National Joint Registry dataset. Bone Joint J. 2015 Aug;97-B(8):1076-81. doi: 10.1302/0301-620X.97B8.35170. PMID 26224824
- [Background] Stelzer W, Aiglesberger M, Stelzer D, Stelzer V. Use of cooled radiofrequency lateral branch neurotomy for the treatment of sacroiliac joint-mediated low back pain: a large case series. Pain Med. 2013 Jan;14(1):29-35. doi: 10.1111/pme.12014. Epub 2012 Dec 28. PMID 23279364
- [Derived] Lyman JR, Olscamp AJ, Lovell TP, Winegar CD, Wilson AN. Radiofrequency ablation prior to total knee arthroplasty does not improve post-surgical pain or recovery: a double-blinded, multi-center, randomized clinical trial. Ann Jt. 2023 Jan 15;8:5. doi: 10.21037/aoj-22-33. eCollection 2023. PMID 38529234